CLINICAL TRIAL: NCT02910180
Title: Genetic, Metabolic, and Growth Factor Repository for Cerebrovascular Disorders
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Nestor R. Gonzalez, MD, MSCR., Professor of Neurosurgery, Cedars-Sinai Medical Center
Other Study IDs: Pro00045392
Record Dates: First submitted 2016-09-14; First posted 2016-09-21 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cerebrovascular Diseases; Ischemic Stroke; Repository
Keywords: Tissue Repository; Cerebrovascular Diseases; Stroke; Aneurysm; Arteriovenous malformation; Fistula; Intracranial Stenosis; Treatment; Registry; Outcomes
MeSH Terms: conditions — Cerebrovascular Disorders; Ischemic Stroke; Stroke; Aneurysm; Arteriovenous Malformations; Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood samples, microdialysis samples, cerebral spinal fluid, and tissue.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Repository Group: The Repository Group consists of patients which have donated tissue to the repository.

SUMMARY:
This study encompasses the maintenance and utilization of a repository of samples from patients with cerebrovascular disease and stroke. The types of tissue taken are blood, cerebrospinal fluid (CSF), tissue, and microdialysis samples. Future analysis of these samples can potentially help investigators to better categorize groups of patients, understand the underlying etiology of these pathologies, identify markers that are associated with favorable or poor outcomes, and track changes that occur during the natural course of the disease or with treatment. This is a prospective observational study which will use samples from such patients to create this library which can be used to explore these questions in the future.

DETAILED DESCRIPTION:
Genetic and metabolic profiling has become an important means to evaluate various pathologies, their effects on patients, and their treatments. In regards to cerebrovascular disease and stroke, there are a number of hypotheses which have been proposed. The levels and types of various angiogenic factors in the blood and tissues have been proposed to be predictive of patient outcome after ischemic stroke and treatment for stroke. Likewise, genetic factors may predict outcome or response to various types of treatments.

The role of biological samples in furthering our understandings about cerebrovascular disease and treatment are well documented. Muscle microdialysis samples have confirmed the presence of sublethal ischemia during the induction of remote ischemic preconditioning. The effects of remote ischemic preconditioning on the coagulation profile, DNA methylation, and cell cycle gene expression of patients with aneurysmal subarachnoid hemorrhage have also been elucidated. Blood samples collected in patients with intracranial arterial stenosis have produced many insights. Inflammatory cell profiles in patient who receive encephaloduroarteriosynangiosis (EDAS) surgery have been characterized. Angiogenic factor measurements have been shown to predict the degree of neovascularization in patients post-EDAS. In patients with intracranial atherosclerosis, angiogenic factor profiles were found to strongly correlate with failure of medical management and poor outcomes.

It is clear that genetic and metabolic profiling are effective tools in evaluating the effects of cerebrovascular disease and their treatments. This study encompasses the maintenance and utilization of a repository of samples from patients with cerebrovascular disease and stroke. For every patient enrolled in the study, relevant patient information such as age, gender, diagnosis, medical history, family history, procedures/treatments received, radiological reports, and patient outcomes are recorded. This information is updated upon every follow-up during the study. The types of tissue taken are blood, cerebrospinal fluid (CSF), tissue, and microdialysis samples.

Future analysis of these samples can potentially help investigators to better categorize groups of patients, understand the underlying etiology of these pathologies, identify markers that are associated with favorable or poor outcomes, and track changes that occur during the natural course of the disease or with treatment. This repository serves as the groundwork to explore these questions in the future.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with cerebral vascular disease, regardless of gender, age, ethnicity/race, stage of disease or treatment, are eligible.
* Expected availability of clinical follow up data
* Participants must be willing to provide written, informed consent obtained in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Pregnant women are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with cerebrovascular disease. This includes both non-surgical patients (such medically managed ischemic stroke, aneurysms, moyamoya disease, arteriovenous malformation, hemorrhagic stroke, etc.) and surgically treated patients (patients with aneurysm coiling or clipping, arteriovenous malformation resection, direct or indirect revascularization procedures for ischemia, etc.).
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2016-09; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in modified Rankin Scale (mRS) score | Baseline, 1 Month, 3 Months, and 6 Months
Change in NIH Stroke Scale score | Baseline, 1 Month, 3 Months, and 6 Months
Change in Barthel Index | Baseline, 1 Month, 3 Months, and 6 Months
Change in Montreal Cognitive Assessment test score | Baseline, 1 Month, 3 Months, and 6 Months

SECONDARY OUTCOMES:
Change in Angiographic Neovascularization | Baseline and 6 Months
  Analyzed in digital subtraction angiography (DSA) images
Change in Angiogenic Factor Measurements | Baseline, 1 Month, 3 Months, 6 Months
  Measured in blood, CSF, microdialysis samples, and tissue

CONTACTS AND LOCATIONS:
Overall Officials: Nestor R Gonzalez, MD, MSCR, Principal Investigator — Cedars-Sinai Neurosurgery
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Mayor F, Bilgin-Freiert A, Connolly M, Katsnelson M, Dusick JR, Vespa P, Koch S, Gonzalez NR. Effects of remote ischemic preconditioning on the coagulation profile of patients with aneurysmal subarachnoid hemorrhage: a case-control study. Neurosurgery. 2013 Nov;73(5):808-15; discussion 815. doi: 10.1227/NEU.0000000000000098. PMID 23867300
- [Background] Nikkola E, Laiwalla A, Ko A, Alvarez M, Connolly M, Ooi YC, Hsu W, Bui A, Pajukanta P, Gonzalez NR. Remote Ischemic Conditioning Alters Methylation and Expression of Cell Cycle Genes in Aneurysmal Subarachnoid Hemorrhage. Stroke. 2015 Sep;46(9):2445-51. doi: 10.1161/STROKEAHA.115.009618. Epub 2015 Aug 6. PMID 26251247
- [Background] Ooi YC, Laiwalla AN, Liou R, Gonzalez NR. Angiographic Structural Differentiation between Native Arteriogenesis and Therapeutic Synangiosis in Intracranial Arterial Steno-Occlusive Disease. AJNR Am J Neuroradiol. 2016 Jun;37(6):1086-91. doi: 10.3174/ajnr.A4675. Epub 2016 Jan 21. PMID 26797139
- [Background] Bilgin-Freiert A, Dusick JR, Stein NR, Etchepare M, Vespa P, Gonzalez NR. Muscle microdialysis to confirm sublethal ischemia in the induction of remote ischemic preconditioning. Transl Stroke Res. 2012 Jun;3(2):266-72. doi: 10.1007/s12975-012-0153-1. Epub 2012 Apr 10. PMID 24323782
- [Background] Dusick J, Hamilton R, Bilgin-Freiert A, Vespa P, Hu X, Asgari S, Gonzalez NR. Immediate Cerebrovascular and Brain Metabolic Effects of Remote Ischemic Preconditioning. Stroke; a journal of cerebral circulation. 2012; 43:A2698.
- [Background] Gonzalez, N. R., Liou, R. J., Rao, N., Hinman, J. D., Restrepo, L., Ali, L., … Saver, J. (2016). Abstract TP119: Angiogenic Factor Profiling in Medical Treatment of Intracranial Atherosclerosis (ICAS). Stroke, 47(Suppl 1), ATP119-ATP119.
- [Background] Gonzalez, N. R., Ooi, Y., Laiwalla, A., Restrepo, L., Ali, L., Liou, R., … Saver, J. (2016). Abstract TMP15: Circulating Antiangiogenic Profile Predicts Lower Degrees of Neovascularization After Indirect Revascularization With Encephaloduroarteriosynangiosis (EDAS) in Patients With Intracranial Atherosclerosis (ICAS). Stroke, 47(Suppl 1), ATMP15-ATMP15.
- [Background] Gonzalez, N. R., Connolly, M. J., Ooi, Y. C., Dusick, J., Bounni, F., Liebeskind, D. S., … Iruela-Arispe, L. (2015). Abstract 135: Angiogenic Factors and Response to Intensive Medical Management in Atherosclerotic Intracranial Arterial Stenosis. Stroke, 46(Suppl 1), A135-A135.
- [Background] Gonzalez, N. R., & Iruela-Arispe, L. (2014). Abstract T P90: Characterization of Inflammatory Cells after EDAS Surgery in Patients with Intracranial Arterial Stenosis. Stroke, 45(Suppl 1), ATP90-ATP90.
- [Background] Gonzalez, N. R., Liou, R., Ooi, Y., Hinman, J. D., Rao, N., Toscano, J., … Saver, J. (2016). Abstract WP138: Effects of Intensive Medical Management (IMM) and Encephaloduroarteriosynangiosis (EDAS) On VEGFA165a/b Ratios in Patients With Intracranial Atherosclerosis (ICASi. Stroke, 47(Suppl 1), AWP138-AWP138.